CLINICAL TRIAL: NCT01091922
Title: Prebiotic Evaluation of Cocoa-derived Flavanols in Healthy Humans Using a Randomized, Double Blind, Crossover, Placebo-controlled Intervention Study
Brief Title: The Impact of Dietary Flavanols on the Gut Microflora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Dr Jeremy P E Spencer, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UReading-2009-01
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Intestinal Bacteria Growth
Keywords: flavonoids; flavanols; bacteria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Flavanol (Placebo Comparator): Low flavanol drink containing 23 mg of total flavanols. Macro- and micro-nutrient matched with active comparator
  Interventions: Dietary Supplement: Low flavanol cocoa beverage
- High Flavanols (Active Comparator): High Flavanol drink containing 495 mg of total flavanols
  Interventions: Dietary Supplement: High flavanol cocoa beverage

INTERVENTIONS:
Dietary Supplement: Low flavanol cocoa beverage — 23 mg of total flavanols from cocoa
  Arms: Low Flavanol
Dietary Supplement: High flavanol cocoa beverage — 495 mg of total flavanols from cocoa
  Arms: High Flavanols

SUMMARY:
The primary propose of this study is to determine the impact of flavanol-rich cocoa on the growth of the human gut microbiota.

DETAILED DESCRIPTION:
A randomised, placebo-controlled, double-blind, cross-over human intervention study will be conducted in 20 healthy human volunteers to test the impact of a high-flavanol containing meal on the growth of the large intestinal bacteria (microflora). The high flavanol test meal will contain 495 mg of flavanols and the low flavanol control will contain 23 mg of flavanols. The two intervention diets are otherwise matched for macro- and micronutrient content. Changes in the gut microbiota will be determined by measuring bacterial population levels in human faecal material using 16S rRNA targeted oligonucleotide probes and fluorescence in situ hybridization. A number of other biochemical and physiological measures will be recorded including blood glucose, lipoproteins, cytokine levels and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* a signed consent form
* age of 18-50 years inclusive
* BMI between 20-26

Exclusion Criteria:

* pregnant or lactating
* allergy to milk products
* sensitivity to alkaloids and/or caffeine
* gastrointestinal disorders (e.g., chronic constipation, diarrhoea, inflammatory bowel disease, -inflammatory bowel syndrome, or other chronic gastrointestinal complaints)
* diabetes mellitus
* hypertension (>150/90 mm/Hg)
* anaemia and gall bladder problems
* not consuming probiotics, prebiotics, antibiotics or anti-inflammatory or blood lowering medication within a 2-month period prior to the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Faecal bacteria numbers using 16S rRNA targeted oligonucleotide probes analysis and fluorescence in situ hybridization | baseline and 4 weeks
  Measurements of the growth rate and number of bacterial species in human faecal samples using 16S rRNA targeted oligonucleotide probes and fluorescence in situ hybridisation.

SECONDARY OUTCOMES:
Blood pressure | Baseline, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Spencer, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Tzounis X, Rodriguez-Mateos A, Vulevic J, Gibson GR, Kwik-Uribe C, Spencer JP. Prebiotic evaluation of cocoa-derived flavanols in healthy humans by using a randomized, controlled, double-blind, crossover intervention study. Am J Clin Nutr. 2011 Jan;93(1):62-72. doi: 10.3945/ajcn.110.000075. Epub 2010 Nov 10. PMID 21068351